CLINICAL TRIAL: NCT04063722
Title: A Randomized Controlled Trial Modified Benelli Procedure For Subcutaneous Mastectomy In Gynecomastia
Brief Title: Modified Benelli Procedure For Subcutaneous Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7 Al-KindyCM
Record Dates: First submitted 2019-07-30; First posted 2019-08-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2019-08

CONDITIONS: Gynecomastia; Surgical Incision
MeSH Terms: conditions — Gynecomastia; Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Benelli Procedure (Experimental): point x refers to the point where the nipple areola complex should be placed at 18 cm from the mid clavicular line. line A is marked above and medial to the areola and a second radial line above it and parallel to it passing in the point (X) was made and named line B. The ends of this line is curved to approximate and connect to both ends of the line A . two incisions were made on the lines A and B . Next, the whole thickness of the excess skin between line A and the line B was excised (Simon classification 2A, 2B and 3) and subcutaneous mastectomy was done and sent to histopathology. Later on, bleeding control was done by good hemostasis and suction drain was put in its proper site. Finally subcuticular suturing was done by approximation of two incisions using Nylon 3/0. Lastly, sterile pressure dressing was placed.
  Interventions: Procedure: modified Benelli procedure
- webester procedure (Active Comparator): periareolar incision with excision of the breast tissue
  Interventions: Procedure: modified Benelli procedure

INTERVENTIONS:
Procedure: modified Benelli procedure — use of modified Benelli procedure for surgical treatment of gynecomastia

SUMMARY:
The study included 150 patients with gynecomastia (Grade II and III) for the period between January 2010 and January 2016 who attended private hospitals and Al- Kindy Teaching Hospital. The patients were divided into two groups according to the operative techniques used. Group A included 75 patients treated surgically with subcutaneous mastectomy using periareolar incision. Group B; included the other 75 patients who were managed by "modified Benelli technique". The subcutaneous mastectomy using "modified Benelli technique" showed a significantly lower operating time due to ample access for excision of breast tissue. Excision of excess skin allowed the areola to retain a cosmetically more acceptable position. There was a lot of pleating of the skin compared to the other technique using the periareolar incision.

DETAILED DESCRIPTION:
Patients with true gynecomastia, attending Al-Kindy Teaching Hospital and private hospitals, Baghdad, Iraq, from January 2010 to January 2016 were enrolled in the study. Grading of gynecomastia was done according to Cordova and Moschella classification (6). Patients with Grade I were excluded because of no skin excess, while grade IV were excluded due to the need of more extensive procedures. The study protocol was reviewed and approved by the Scientific and Ethical Committee of Al-Kindy College of medicine and Al-kindy Teaching hospital in the committee number 6 in 20-5-2019 (Ethical approval number and Date). Written informed consents were obtained from all patients as an action on acceptance. All enrolled patients were operated by the same surgeon. Patients were randomly assigned to one of the following surgical technique: Group A; included patients who underwent subcutaneous mastectomy using periareolar incision with lateral and medial extension as needed according to Webster(12).

Group B; included patients who were treated by the proposed Modified Benelli Technique (MBT) using the following operative procedure:

First ask the patient to stand up and draw the a line referring to the midline of the chest then mark the ideal breast meridian at 18 cm from midclavicular point to show the position where the nipple should be placed (point X) with skin marker pen and assess the quantity of surplus skin to be excised. After that, ask the patient to lie down on the couch and a periareolar line was marked ( line A) above and medial to the areola and a second radial line above it and parallel to it passing in the point (X) was made and named line B. The ends of this line is curved to approximate and connect to both ends of the line A . Then, the patient is given general anesthesia and the two incisions were made on the lines A and B i.e. periareolar incision above and medial to the areola with a second incision above it and connecting both ends . Next, the whole thickness of the excess skin between line A and the line B was excised (Simon classification 2A, 2B and 3) and subcutaneous mastectomy was done and sent to histopathology. Later on, bleeding control was done by good hemostasis and suction drain was put in its proper site. Finally subcuticular suturing was done by approximation of two incisions using Nylon 3/0. Lastly, sterile pressure dressing was placed. The result of both groups were compared in terms of operating time, nipple-areola complex location, post-operative complications including, pleating of the skin at suture line, hematoma, bruising at the site of incision, , soft tissue deformity, seroma, hypoesthesia of nipple-areola complex, wound dehiscence, areolar epidermolysis, and hypertrophic scarring.

ELIGIBILITY:
Inclusion Criteria:

* all patients with gynecomastia

Exclusion Criteria:

* Patients with Grade I gynecomastia because of no skin excess
* patients with grade IV due to the need of more extensive procedures

Ages: 17 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
prevalence of proper postoperative nipple-areolar complex position: the distance from the midclavicular point to the postoperative nipple areola complex position. | Documented on one occasion, at 6 months postoperatively.
  The distance from the midclavicular point to the nipple areola complex position were measured postoperatively, with an average of 6-month follow-up, to evaluate the aesthetic appropriateness of the postoperative nipple areola complex position which should be 18-19 cm from the midclavicular point.

CONTACTS AND LOCATIONS:
Overall Officials: Riyadh M Hasan, C.A.B.S., Study Chair — Al kindy college of medicine university of Baghdad